CLINICAL TRIAL: NCT06347939
Title: Mediastinal Endobronchial Ultrasound Bronchoscopy Cryobiopsy Study In Sweden
Brief Title: Mediastinal EBUS Cryobiopsy Study In Sweden
Acronym: MECRIS
Status: Recruiting | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Hamid Akbarshahi, Pulmonary medicine specialist, Region Skane
Other Study IDs: 2023-06638-01
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-06

CONDITIONS: Mediastinal Lymphadenopathy; Lung Cancer; Sarcoidosis; Lymphoma; Tuberculosis
Keywords: Mediastinal lymphadenopathy; Lung cancer; Sarcoidosis; Tuberculosis; Lymphoma
MeSH Terms: conditions — Lung Neoplasms; Sarcoidosis; Lymphoma; Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Lymph node biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All the patients undergo the same procedure: All the patients undergo the same procedure and every patient's own samples are compared to each other.
  Interventions: Diagnostic Test: Mediastinal lymph nodes cryobiopsies

INTERVENTIONS:
Diagnostic Test: Mediastinal lymph nodes cryobiopsies — EBUS Mediastinal lymph nodes cryobiopsies
  Other Names: Mediastinal lymph nodes fine needle aspiration

SUMMARY:
This study is a prospective observational non-randomized clinical trial where all the participitants undergo the same procedure and every participitant's samples are compared to each other. The investigators conduct EBUS TBNA and EBUS TBMCB on all the study participants.The cryobiopsy samples are numbered to evaluate the number of biopsies needed to reach a definite diagnosis and to assess the added value of every sample taken from the same participitant. Every participitant's own samples are compared to each other and added value of EBUS TBMCB is defined as the difference in diagnostic yield between the EBUS TBNA alone and the combination of EBUS TBNA with EBUS TBMCB. Diagnostic yield is defined as the efficacy of the investigation module in reaching a definite diagnosis (percentage of cases with a definite diagnosis).

Follow up four weeks after the procedure to assess the risk for postoperative complications.

DETAILED DESCRIPTION:
Endobronchial ultrasound bronchoscopy (EBUS) is an established method for sampling of mediastinal and hilar lymph nodes and masses. Cytology specimens can be obtained with transbronchial needle aspiration (EBUS TBNA), and this is a valuable tool in the diagnostic work up of lesions adjacent to central airways and in the staging of lung cancer. EBUS TBNA is a robust method that shows excellent results in diagnosing lung cancer cases with a reported diagnostic yield up to 90% from multiple studies. EBUS TBNA is a safe procedure with reported complications in 1,2 - 3,6% of cases.

In clinical situations where non-malignant diseases (e.g. sarcoidosis, tuberculosis) or malignancies other than lung cancer (e.g. lymphoma) affect the mediastinum is the efficacy of EBUS TBNA relatively limited and these cases often require histopathological evaluation rather than cytological assessment.

EBUS TBMCB (EndoBronchial UltraSound TransBronchial Mediastinal CryoBiopsy) is a novel method of obtaining cryobiopsies for histopathology from mediastinal lesions, which has previously not been possible with endobronchial procedures. This method is becoming more utilised internationally after the publication of the first studies examining its safety and efficacy. In the last couple of years has EBUS TBMCB been evaluated in two randomized studies from the same study group and a few observational studies where adding EBUS TBMCB to EBUS TBNA showed an increase in diagnostic yield without adding significant adverse events. The sensitivity of EBUS TBMCB were similar to that of EBUS TBNA in cases of lung cancer but there was found, in all studies, a significant increase of diagnostic yield in cases of non-malignant diseases and metastases from extra thoracic tumours.

There are however some aspects of this novel method yet not studied like the number of biopsies needed from a lesion to collect adequate material for histopathological evaluation. At the thoracic oncology diagnostics units at Skåne University Hospital and Umeå University hospital, EBUS TBMCB has been introduced in clinical practice, performed by experienced bronchoscopists. In recognition of the need for further clarification regarding several aspects of this novel method the investigators plan to collect data prospectively and systematically from EBUS TBMCB procedures.

Our study is a prospective observational non-randomized clinical trial where all the patients undergo the same procedure and every patient's own samples are compared to each other. The investigators conduct EBUS TBNA and EBUS TBMCB to all the study participants and the investigators are numbering the cryobiopsy samples to evaluate the number of biopsies needed to reach a definite diagnosis and to assess the added value of every sample taken from the same patient. Every participitant's own samples are compared to each other and added value of EBUS TBMCB is defined as the difference in diagnostic yield between the EBUS TBNA alone and the combination of EBUS TBNA with EBUS TBMCB. Diagnostic yield is defined as the efficacy of the investigation module in reaching a definite diagnosis (percentage of cases with a definite diagnosis).

Follow up four weeks after the procedure to assess the risk for postoperative complications.

Data will be collected in both sites from all EBUS TBMCB procedures eligible according to inclusion criteria, where patients agree to partake in the study, until 200 cases are reached.

ELIGIBILITY:
Inclusion Criteria:

* Mediastinal lymphadenopathy with a diameter greater than 1 cm.
* Indication for assessment and sampling according to clinical praxis
* Age > 18 years
* Patients consent to participate in the study.

Exclusion Criteria:

* Hemodynamically instable patient
* Myocardial infarction in the last six weeks prior to participating in the study.
* Life threatening arrythmia
* Respiratory failure and inadequate blood oxygenation despite oxygen supply.
* Tracheal obstruction of high grade.
* High bleeding risk
* Patient not willing to participate in the study
* Patient not speaking swedish and needing translator during the procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years with mediastinal lymphadenopathy with a diameter greater than 1 cm who have indication to undergo sampling of lymph nodes for assessment according to clinical praxis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of mediastinal cryobiopsies needed per patient to lead to a definite diagnosis. | 2 years
  The result will be presented as the mean value of the number of biopsies needed to analyze for each individual to reach a definite diagnosis.

SECONDARY OUTCOMES:
Adequacy of mediastinal cryobiopsies for PDL1 analysis in lung cancer. | 2 years
  Material leading to a definite answer is considered adequate.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Respiratory medicine and allergy department, Skåne University Hospital, Lund
  - Norrlands universitetssjukhus, Umeå